CLINICAL TRIAL: NCT02864459
Title: The Role of Muscular Ultrasound in Predicting Weaning Success
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jinwoo Lee, Associate professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 690
Record Dates: First submitted 2016-08-07; First posted 2016-08-12 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Respiratory Insufficiency
Keywords: Ultrasonography; Weaning
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Muscular ultrasound (Experimental)
  Interventions: Other: Muscular ultrasound

INTERVENTIONS:
Other: Muscular ultrasound — Muscular ultrasound is done before extubation

SUMMARY:
When attempting to wean a patient from the ventilator, even if he/she passes the spontaneous breathing test, 10-20% of the time extubation failure occurs and the patient is reintubated. When the patient is reintubated the mortality rate increases and the length of intensive care unit stay is also increased. It is vital to intensively assess the patient before extubation and correctly predict extubation success. Muscular ultrasound may be helpful in these situations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing weaning from mechanical ventilation
* Patients who have been mechanically ventilated for more than 72 hrs

Exclusion Criteria:

* Pregnant patients
* Patients with previous neuromuscular diseases
* Difficulties in muscular ultrasound (Dressing, operation, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2016-08; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Extubation success (no need for reintubation) | 48 hours after extubation

SECONDARY OUTCOMES:
Weaning success (no need for applying the ventilator again) | 2 hours after spontaneous breathing trial

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided